CLINICAL TRIAL: NCT05529979
Title: Post-Market Clinical Follow-Up Study of a Robotic Device for Image Guided Percutaneous Needle Placement in the Abdomen
Brief Title: Epione® Post-Market Clinical Follow-up Study
Acronym: SaFE
Status: Completed | Type: Observational
Sponsor: Quantum Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: QS-NIS-G-H-2101
Record Dates: First submitted 2022-06-07; First posted 2022-09-07 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-08

CONDITIONS: Cancer Abdomen
Keywords: Percutaneous; CT-guided; Ablation; Biopsy; Abscess Drainage; Fiducial Placement; Abdomen; Liver; Kidney; Robotics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Intervention with the EPIONE® device: Patients treated by percutaneous CT-guided procedures in the abdomen with the EPIONE® device
  Interventions: Device: EPIONE® CT-Guided Percutaneous procedures

INTERVENTIONS:
Device: EPIONE® CT-Guided Percutaneous procedures — The EPIONE device is a user controlled, stereotactic accessory intended to assist in the planning and manual advancement of one or more instruments, as well as in verification of instrument position during Computed Tomography (CT) guided percutaneous procedures.

SUMMARY:
Post-Market Clinical Follow-up study in order to consolidate performance and safety data of the EPIONE® device when used for percutaneous procedures in the abdomen

DETAILED DESCRIPTION:
The objective of this PMCF study is to compile data on the routine use of the EPIONE® device in subjects undergoing CT-guided percutaneous procedures in the abdomen.

The objectives are:

1. to evaluate the technical success of the device
2. to evaluate performance parameters (accuracy measures, adjustements, post-intervention ablation success, local tumor recurrence, operator satisfaction) and the safety of the device

55 patients are planned in this post-market study.

ELIGIBILITY:
Inclusion Criteria:

* Patient >18 years old,
* Patient for whom a CT-guided procedure in abdomen has been prescribed and agreed by a multidisciplinary team of radiologists, surgeons and clinicians,
* Patient with a confirmed non-opposition.

Exclusion Criteria:

* Patient unable to undergo general anesthesia,
* Pregnant or breast-feeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated/operated in routine practice, in accordance with the device's intended use, without any additional nor burdensome procedure.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2024-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Baptiste BONNET, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy Institut, Villejuif, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 55 patients were included (28-Apr-2022 and 20-Jan-2023) at the IGR (Villejuif/France). The date of the last patient FU visit is 27-APR-2024.
Units Other Than Participants: tumor lesions
Period: Overall Study
Arm/Group | Intervention With the EPIONE® Device
Started | 55; 62 tumor lesions
Completed | 40; 56 tumor lesions
Not Completed | 15; 6 tumor lesions
Not completed — Lost to Follow-up | 6
Not completed — Physician Decision | 1
Not completed — non-feasibility cases | 4
Not completed — Lack of Efficacy | 3
Not completed — ablation not performed | 1

BASELINE CHARACTERISTICS:
Population: 55 patients were included but 54 were analysed (1 patient was registered under 2 inclusion n°: n°3 and n°55. Patient n°55 was included due to tumor recurrence but was subsequently withdrawn from the study after consultation with the principal investigator, as the protocol does not account for the evaluation of secondary efficacy outcomes).
  Among the 54 patients analysed: 30 males (55.6%) and 24 females (44.4%) representing 61 lesions which required 108 needle insertions during 56 procedures.
Arm/Group | Intervention With the EPIONE® Device
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 54

OUTCOME MEASURES:

1. Primary Outcome: Technical Success
Description: Number of targets reached ; the target is considered to have been reached when the needle is positioned accurately enough to allow the planned procedure to be performed (by patient)
Time Frame: Visit 2 - D0 The day of the intervention
Population: The Screened, ITT, PP and Safety populations were identical, each comprising 54 patients
Measure: Number; unit: Participants
Arm/Group | Intervention With the EPIONE® Device
Number analyzed (Participants) | 54
Participants | 50

2. Primary Outcome: Technical Success
Description: Number of targets reached ; the target is considered to have been reached when the needle is positioned accurately enough to allow the planned procedure to be performed (by lesion)
Time Frame: Visit 2 - D0 The day of the intervention
Population: The Screened, ITT, PP and Safety populations were identical, each comprising 61 lesions.
Measure: Number; unit: lesions
Units Other Than Participants: Lesions
Groups:
- Intervention With the EPIONE® Device: Lesions treated by percutaneous CT-guided procedures in the abdomen with the EPIONE® device
  EPIONE® CT-Guided Percutaneous procedures: The EPIONE device is a user controlled, stereotactic accessory intended to assist in the planning and manual advancement of one or more instruments, as well as in verification of instrument position during Computed Tomography (CT) guided percutaneous procedures.
Arm/Group | Intervention With the EPIONE® Device
Number analyzed (Participants) | 54
Number analyzed (Lesions) | 61
lesions | 56

3. Secondary Outcome: Needle Placement Accuracy
Description: accuracy of the needle placement: deviation between the planned and actual needle position once inserted
Time Frame: Visit 2 - D0 The day of the intervention
Reporting Status: Not Posted

4. Secondary Outcome: Number and Nature of Needle Adjustments to Reach the Target
Description: Detail of the number/nature of adjustments performed after the initial insertion of the needle
Time Frame: Visit 2 - D0 The day of the intervention
Reporting Status: Not Posted

5. Secondary Outcome: Post-intervention Ablation Success
Description: Minimal Ablation Margin(s) measure(s) if applicable (mm)
Time Frame: Until Visit 4 - Routine FU visit at 10 months
Reporting Status: Not Posted

6. Secondary Outcome: Local Tumor Recurrence
Description: Evaluation of the local tumor progression following the ablation (if applicable)
Time Frame: Until Visit 4 - Routine FU visit at 10 months
Reporting Status: Not Posted

7. Secondary Outcome: Operator Satisfaction
Description: 5-point Likert scale: very Dissatisfied/dissatisfied/neutral/satisfied/highly satisfied
Time Frame: Visit 2 - D0 The day of the intervention
Reporting Status: Not Posted

8. Secondary Outcome: Adverse Events Related to Device or Procedure
Description: Safety of the device
Time Frame: Until Visit 4 - Routine FU visit at 10 months
Reporting Status: Not Posted

9. Secondary Outcome: Device Dysfunction
Description: Evaluation of the device dysfunction
Time Frame: Visit 2 - D0 The day of the intervention
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The safety population is composed of the 54 included patients who were followed until 2 months (88.9% of patients) and 10 months (72,2% of patients).
Description: Intensity, Category, Action, Causality, outcome, patient and procedural risk modifier, adverse event preventability and management of each adverse event were classified according to SIR classification (Khalilzadeh and al.2017 / Sacks and al.2003). The adverse event category (serious or not) was from the ISO 14155-1.
Arm/Group | Intervention With the EPIONE® Device
All-Cause Mortality (participants affected / at risk) | 0/54
Serious Adverse Events (participants affected / at risk) | 3/54
Other Adverse Events (participants affected / at risk) | 4/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention With the EPIONE® Device (N=54)
Polynephritis requiring prolonged hospitalization (Renal and urinary disorders) | 1 (1)
Hospitalization for large abscess in the thermoablation area, requiring drainage (Infections and infestations) | 1 (1)
Hemorrhagic pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention With the EPIONE® Device (N=54)
Adjacent structure thermal lesion (Surgical and medical procedures) | 1 (1)
Fever (Surgical and medical procedures) | 2 (2)
Pneumothorax with drainage (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
From the protocol:

"Prior to submitting the results of this study for publication or presentation, the Investigator will allow the Sponsor 30 days in which to review and comment upon the publication manuscript. The Sponsor agrees that before he publishes any results of this study, he shall provide the Investigators at least 30 days for full review of the publication manuscript"

DOCUMENTS (2):
  • Study Protocol (2022-10-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT05529979/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/79/NCT05529979/SAP_001.pdf